CLINICAL TRIAL: NCT06901193
Title: A Virtual Reality Mindfulness-based Intervention: The Impact and Acceptability for Nurse Managers in an Academic Medical Center
Brief Title: A Virtual Reality Mindfulness-based Intervention for Nurse Managers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Beth Steinberg, Associate Director of Research, Ohio State University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024B0251
Record Dates: First submitted 2025-03-03; First posted 2025-03-28 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-02

CONDITIONS: Perceived Stress; Burnout; Resilience, Psychological; Work Engagement
Keywords: mindfulness; virtual reality; nurse; nurse manager
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Intervention, wait-list control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Participation in the virtual reality mindfulness intervention the first 8 weeks
  Interventions: Behavioral: Virtual Reality Mindfulness intervention
- Wait-list control group (Active Comparator): will participate in the virtual reality mindfulness intervention during the second 8 weeks of the study
  Interventions: Behavioral: Virtual Reality Mindfulness intervention

INTERVENTIONS:
Behavioral: Virtual Reality Mindfulness intervention — Mindfulness will be offered via a virtual reality headset; participants will use the virtual reality mindfulness program 3 times per week (15 minutes at a time) for 8 weeks.

SUMMARY:
A pilot intervention wait-list control study evaluating the effectiveness of a worksite, on-demand virtual reality mindfulness intervention. Outcomes of interest include perceived stress, burnout, work engagement, resilience and respiratory rates. System usability of the VR mindfulness program and integration into the clinical workday will also be assessed for both groups.

DETAILED DESCRIPTION:
This pilot intervention waitlist control study will evaluate the effectiveness of an 8-week on-demand worksite virtual reality mindfulness-based intervention with academic medical center nurse managers and assistant nurse managers. Individual outcome measures will include perceived stress, burnout, resilience, work engagement, weekly respiratory rates, system usability and integration of the intervention into the workday. The study will use a convenience sample of nurse managers and assistant nurse managers recruited from across The Ohio State University Wexner Medical Center. All participants will provide informed consent which will describe the intervention and wait list control groups, the intervention, and the intervention timelines per requirements of the institutional Internal Review Board. After randomization into intervention and waitlist control groups, all participants will complete outcome measures at the same time one week before the initiation of the VR intervention group, one week after the last day of the VR intervention for the intervention group, and again one week after the waitlist control group receives the VR intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Employed as a Nurse Manager or Assistant Nurse Manager at The Ohio State University Wexner Medical Center
* Manage a hospital-based department/unit with supervisory responsibility
* Ability to participate in study for 8 consecutive weeks using VR technology, three times a week for 10-15-minute sessions during work hours

Exclusion Criteria:

* Less than 18 years of age
* Pregnant
* Not employed as a Nurse Manager or Assistant Nurse Manager at The Ohio State University Wexner Medical Center
* Inability to participate in study for 8 consecutive weeks using VR technology, three times a week for 15-minute sessions during work hours.
* Does not have a personal smart phone or computer to access app.
* Inability to read and/or understand English (consent and questionnaires in English)
* Medical or other conditions that would preclude use of Virtual Reality technology such as:
* Epilepsy or neurological conditions where visual stimuli may trigger seizures or other issues, sensitivity to light or motion, current pregnancy, or any injuries that would prevent operating a headset, history of motion sickness or nausea, history of migraines or headaches, history of balance issues or dizziness, pregnancy, recent concussions, or other conditions where dizziness, nausea or headaches are more likely
* Any exclusions determined from the VR Prescreening Questionnaire for Pre-existing Conditions or Prescreening Eligibility Questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-07-12 (Actual); Study Completion 2025-07-12 (Actual)

PRIMARY OUTCOMES:
Perceived Stress | Baseline and on completion of the 8-week intervention
  Perceived Stress Scale-10 (PSS-10). A 10-item self-report measure of perceived stress. It is a measure of the degree to which situations in one's life are appraised as stressful over the past month. The 4-point Likert Scale includes responses of 0 (never), 1 (almost never), 2 (sometimes), 3 (fairly often), and 4 (very often). Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Maslach Burnout Inventory (MBI-HSS) | baseline and on completion of the 8-week intervention
  The MBI-HSS is a self-report assessment of perceptions of burnout specific to healthcare providers. The 22-items describe job-related feelings that healthcare providers may experience in the workplace and encompasses three sub scales of emotional exhaustion, depersonalization, and personal accomplishment. The Likert scale responses include 0 (never), 1 (a few times a year or less), 2 (once a month or less), 3 (a few times a month), 4 (once a week), 5 (a few times a week), and 6 (every day). Each sub scale can have a total score of low, moderate, or high with emotional exhaustion scores: low 0-18, moderate 19-26, high 27 or greater; depersonalization scores: low 0-5, moderate 6-9, high 10 or greater; and personal accomplishment scores: low greater than 40, moderate 34-39, and high 0-33.
Resilience | baseline and on completion of the 8-week intervention
  The Connor-davidson Resilience Scale-10 (CD-RISC-10) is a 10-item self-report assessment of a person's ability to bounce back after adversity. A 5-point Likert Scale for each statement ranges from 0 (Not True at All), 1 (Rarely True), 2 (Sometimes True), 3 (Often True), 4 (True Nearly All of the Time). A respondent's total score can range from 0 to 40 with higher scores indicating higher resilience.
Work engagement | baseline and on completion of the 8-week intervention
  The Utrecht Work Engagement Scale-9 (UWES-9) is a 9-item assessment of attitudes towards one's job. The UWES-9 measures three primary factors including dedication, vigor, and absorption. Each subscale score, answered on a seven-point Likert scale ranging from 0 (Never), 1 (Almost never, a few times a year or less), 2 (Rarely, once a month or less), 3 (Sometimes, a few times a month), 4 (Often, once a week), 5 (Very often, a few times a week), and 6 (Always, every day), has a range of 0 to 18. Higher scores for each sub scale indicate higher dedication, vigor, and absorption with work.
Respiratory rate | The 30-second count of inhalations will be completed by the participant before and after using the virtual reality mindfulness intervention at least three times per week for the entirety of the 8-week intervention
  A self-measured count of inhalations (respiratory rate) taken over a 30-second time period. The participant will place their right hand over their left chest and count inhalations for a 30-second time period before they participate in the virtual reality mindfulness intervention and after they participate in the virtual reality mindfulness intervention.

SECONDARY OUTCOMES:
System Usability Scale | Completed after the 8-week intervention
  The System Usability Scale (SUS) is a 10-item scale measuring usability of a new technology or system. In this study, the SUS will be used to measure the usability of the virtual reality mindfulness intervention. Participants respond to each statement using a 5 point Likert Scale that ranges from 1 (strongly disagree), 2 (disagree), 3 (neither disagree or agree), 4 (agree), and 5 (strongly agree). Total scores range from 0-100 with higher scores indicating higher usability. In general, scores > 80 indicate high usability with scores 50 or less indicating low usability.
Feasibility of Intervention Measure | Participants will complete after completion of the 8-week intervention
  The Feasibility of Intervention Measure (FIM) is a 4-item self-report assessment to evaluate integration of the mindfulness-based intervention into the daily workflow of the nurse manager. Each statement is scored with a 5-point Likert Scale that includes 1 (completely disagree), 2 (disagree), 3 (neither agree nor disagree), 4 (agree), and 5 (completely agree). Total scores range from 4-20 with higher total scores indicating higher feasibility.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD that will be shared will include mean participant age (years) , mean time as a Registered Nurse (years/months), mean time in a Nurse Manager role (years/months), mean number of direct reports, overview of nursing specialities represented in the participant sample, i.e. Medical-Surgical, Intermediate Care, Critical Care, Ambulatory, Other (Peri-op, Obstetrical). In addition, differences in mean pre-intervention and post-intervention scores for intervention and wait-list control groups, significance and effect sizes. De-identified, curated data will be entered into Dryad, an online repository endorsed by The Ohio State University.
Supporting Information: ICF, CSR, Analytic Code
Time Frame: IPD will be available 10-30-2025 and be accessible indefinitely.
Access Criteria: De-identified and curated demographic, statistical data, study overview, study consent will be accessible to academic researchers and educators through a data accessibility link once the Dryad submission is finalized.

REFERENCES:
- Available data/document: Study Protocol — https://orapps.osu.edu/buck-irb/index/view/study/64513